| | THE PERSON NAMED IN | | | | | 6 | THE THE THE TREE THE THE THE THE | Comment. | Ē |
|---|---|---|---|---|---|---|---|---|---|
| į. | Amendment of the same | REPORTED AND AND PARTIES AND ADDRESS OF PRINCIPLES | THE PROPERTY OF THE PROPERTY O | AVERTA AND A STATE OF THE STATE OF | ************************************** | THE THE PERSON NAMED IN COLUMN | | | |
| l | | C | 0 | | | Cill Cill | Sam Dickson | Spensor<br>Representations | ŧ |
| | | enninga | Chaudia Q | 9/18/17 | | mangs. | Chandia Jennous | Spinson Control | 1 |
| أسمده | | £ . | Jan H | 9/13/17 | P | 15.23 | Parithey inc. | Spaniative<br>Repiesemente | |
| | Ø | 5 | 0 | | the day was a second of the se | VIT B IN VANA AND | | WA Moderal Land | ř. |
| | Ø | | | | | - | | HILA Society Level | |
| | Ø | | | | 411700 | Í | | BBA Rogedators | i |
| L | Ø | O. | | -Alle-Tie- | | ************************************** | | BBA Clinical Load | 1 |
| ~~~~~ | | Wood I | 11.47 | 155 Coc- | * | det (Y | Mark Melidaff | B5/2 Sims Lond | 1 |
| <u></u> | | MILLER | | MSEC201 | 100 | CINEST. | Mark Melkluff | Pregrammer Load | |
| | Ø | | | A California de America de California de Cal | Company of the Compan | | | Management Lead | 1 |
| LI | | | 0260 | 1950201 | | | Jane Shaw | SHA Project<br>Manager | 1 |
| | Ø | | | | | | | BBA President | 1 |
| | N/A | leste | Signature | Dare | All the second s | Name | | Functional Role | 7***** |
| 2 | | | | | - | 7. 7. 7 | | COP 71 - L SPAN AMERICA - A ST. CO. CO. C. | |
| <u>, </u> | £ 1000 25 51 | // Date: /9: | White The Boll | ure 2 | Signature | Mark Molldoff | Mark | Document Owner | |
| | SECONDARY OF STREET | Date | | ura. | Signature | | 122 | If Yes, Performed by | |
| | | | AMPLAATI - III OO - III OO - III OO III OO O | No. | M | red Des | ditton Requ | Text and Table Validation Regio ed? | i |
| ŀ | <u> </u> | B week | Descured Version | PRI PLANTA ALABAMAN AND A | SAPI | Statistica: Analysis Papi (SAP) | Statistica | Document Type | |
| | | 05 | Themn RF 005 | Project Title | Pr | *************************************** | ) X [ | Sponsor Therm | |
| Ĺ | A company to the second of the | PAGETOFI | ) Y G | Form | provali | Study Specific Document Review & Approval Form | Documen | Study Specific | F |
| | | æ | REVISION: | | | er e | | A CANADA | |
| | 17.1 | EN GPBUZI | BOT MENT #: | <u></u> | | | | | |
| | | FORM | | <del></del> - | | | | | |
| , | | | Builde to the second of the se | West to the state of the American | ALABAMAT CO. A. A. C. C. | The second second second | of columns of the contrast of | | |

| Study Specific Document Review & Approval Form | BOSTON BIOMEDICAL ASSOCIATES | A PART | |
|---|---|---|---|
| PAGE 1 OF 1 | REVISION: | DOCUMENT #: | FORM |

| | 1 | | | FORM | |
|---|---|---|---|---|---|
| | THE TENTH OF THE T | | DOCUMENT #: | FM GP007.1 | 007.1 |
| | BOSTON IHOMEDICAL ASSO | ASSOCIATES | REVISION: | ET . | |
| Study Specif | Study Specific Document Review & Approval Form | proval Form | Pac | PAGE 1 OF 1 | |
| Sponsor: Thermi | mi | Project Title | Thermi RF 005 | 05 | |
| Document Type: | Statistical Analysis Plan (SAP) | SAP) | Document Version: | rsion: B | |
| Text and Table Va | Text and Table Validation Required? | No. | | | |
| If Yes, Performed by | ву: | Signature: | | Date: | |
| Document Owner: | Mark McIlduff | Signature | | Date: | |
| Functional Role | Name | Date | Signature | ure | N/A |
| BBA President | | | | | |
| BBA Project<br>Manager | Jane Shaw | | | | |
| BBA Data<br>Management Lead | | | | | × |
| BBA SAS<br>Programmer Lead | Mark McIlduff | | | | |
| BBA Stats Lead | Mark McIlduff | | | | |
| BBA Clinical Lead | | | | | × |
| BBA Regulatory Load | | | | | × |
| BBA Safety Lead | | | | | × |
| BBA Medical Lead | | | | | |
| Sponsor<br>Representative | Toni Fournier | | | | |
| Sponsor<br>Representative | Claudia Jennings | | | | |
| Sponsor<br>Representative | Sam Dickson | 1550p 2017 | Sura | | |
| Comments: | | | | | |
| Comments. | | | | | |





# STATISTICAL ANALYSIS PLAN

Protocol Title (Number):

An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental Lift

Thermi\_0005

Sponsor: ThermiGen, LLC

Boston Biomedical Associates 100 Crowley Drive, Suite 216 Marlborough, MA 01752

Effective Date:
SEP 2 0 2017
Initials ΥΝΜΌ Date 1950 2017





#### TABLE OF CONTENTS

| 9 | Baseline Medical History | 8.3 | |
|------|-----------------------------------------------------|--------|-----|
| 9 | Prior and Concurrent Medications | 8.2 | |
| 9 | Demographics | 8.1 | |
| 9 | Demographics and Other Baseline Characteristics | 8 D | |
| 9 | Assessment of Homogeneity | 7.6 | |
| 9 | Multiple Comparisons and Multiplicity | 7.5 | |
| 8 | Protocol Violations | 7.4 | |
| ers8 | Methods for Withdrawals, Missing Data, and Outliers | 7.3 | |
| 8 | Disposition of Subjects and Withdrawals | 7.2 | |
| 8 | Analysis Software | 7.1 | |
| 8 | General Issues for Statistical Analysis | 7 G | |
| 8 | Rater Agreement Population | 6.4 | |
| 7 | Safety | 6.3 | |
| 7 | Per-Protocol Population (PP) | 6.2 | |
| 7 | Intent to Treat Population (ITT) | 6.1 | |
| 7 | Analysis Populations | 6 A | _ |
| 7 | Sample Size | 5 S | |
| 6 | 4.1.3 Safety Endpoints | 4. | |
| 6 | 4.1.2 Secondary Objective/Endpoints | 4 | |
| 6 | 4.1.1 Primary Objective/Endpoint | 4 | |
| 6 | Study Objectives | 4.1 | |
| 6 | Study Objectives and Endpoints | 4<br>S | |
| 6 | Final Analyses and Reporting | 3.2 | |
| 6 | 3.1.2 Other Interim Reports | 3. | |
| 6 | 3.1.1 Annual Reports | 3. | |
| 6 | Interim Analyses | 3.1 | |
| 6 | Sequence of Planned Analyses | S<br>S | 1.5 |
| 5 | Summary | 2<br>S | h > |
| 4 | Abbreviations | 1 A | |





| 8.4 | Screening Physical Exam | 9 |
|---|---|---|
| 9 Treat | Treatment Details | . 9 |
| 10 Efi | nalyses | 10 |
| 10.1 | ss Variable | 10 |
| 10.2 | Secondary Effectiveness Variables | 10 |
| 10.2.1 | Validation of Rater's Assessment | 10 |
| 10.2.2 | Physician – Global Aesthetic Improvement Scale Scores (P-GAIS) | 10 |
| 10.2.3 | 3 Subject – Global Aesthetic Improvement Scale Scores (S-GAIS) | $\Box$ |
| 10.2.4 | 4 Physician – Global Satisfaction Questionnaire (P-GSQ) | $\equiv$ |
| 10.2.5 | Subject – Global Satisfaction Questionnaire (S-GSQ) | $\equiv$ |
| 10.2.6 | 6 Qualitative Assessment Based on 2D Photography | $\equiv$ |
| 10.3 | Exploratory Efficacy Variable - Elasticity | $\equiv$ |
| 11 Sa | Safety Analysis | 12 |
| 11.1 | Numerical Rating Scale (NRS) | 12 |
| 11.2 | All Adverse Events | 12 |
| 11.3 | Adverse Events Leading to Withdrawal | 12 |
| 11.4 | Serious Adverse Events (SAE) | 12 |
| 11.5 | Device or Procedure Related Adverse Events | 12 |
| 11.6 | Deaths | 13 |
| 12 Pla | Planned Subgroup Analyses | 13 |
| 12.1 | Sex. | 13 |
| 12.2 | Age | 13 |
| 12.3 | Per-Protocol | 13 |
| 13 Re | Reporting Conventions | 13 |
| 13.1 | Other Reporting Conventions | 13 |
| Attachmer | Attachment 1. Major Protocol Deviations Evaluability Checklist | 15 |
| Attachmer | Attachment 2. Table, Figure, and Listing Shells | 16 |





#### 1 ABBREVIATIONS

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| AE | Adverse Event |
| BBA | Boston Biomedical Associates |
| CRF | Case Report Forms |
| CSR | Clinical Study Report |
| FDA | United States Food and Drug Administration |
| ITT | Intent-To-Treat Population |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NRS | Numerical Rating Scale |
| P-GAIS | Physician Global Aesthetic Improvement Scale |
| P-GSQ | Physician Global Satisfaction Questionnaire |
| PPP | Per-Protocol Population |
| PRA | Percutaneous Radiofrequency Ablation |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| S-GAIS | Subject Global Aesthetic Improvement Scale |
| S-GSQ | Subject Global Satisfaction Questionnaire |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TEAE | Treatment Emergent AEs |





#### 2 SUMMARY

| TITLE | An open-label, single-center, single-treatment, safety and effectiveness evaluation of percutaneous radiofrequency in achieving submental lift |
|---|---|
| PREFACE | This Statistical Analysis Plan (SAP) describes the planned analysis and reporting for ThermiGen, LLC protocol Thermi_0005 (An open-label, single-center, single-treatment, safety and effectiveness evaluation of percutaneous radiofrequency in achieving submental lift). This study is being conducted to assess the safety and effectiveness of the ThermiRF in the treatment of submental skin laxity. The following documents were reviewed in preparation of this SAP: • Clinical Research Protocol Thermi_0005, issued 10MAY2016 |
| | Case report forms (CRFs) issued 18AUG2016 for Protocol Thermi 0005 |
| PURPOSE | The purpose of this SAP is to outline the planned analyses in support of the Clinical Study Report (CSR) for protocol Thermi_0005. Exploratory analyses not necessarily identified in this SAP may be performed to support the clinical development program. Any post-hoc, or unplanned, analyses not identified in this SAP will be clearly identified in the respective CSR. |
| STUDY<br>OBJECTIVES | The objective of this study is to assess the improvement in overall lift of the submental area at 90 days as determined by a quantitative assessment based on 3D photography. |
| | <b>Primary Efficacy:</b> The primary efficacy endpoint is the improvement in overall lift of the submental area at 90 days as determined by a quantitative assessment based on 3D photography. |
| ENDPOINTS | Secondary Efficacy: The secondary endpoint is overall aesthetic improvement of the submental area and jawline definition at Days 90 and 180 evaluated by the investigator and subject using the following subjective assessments: 1. Qualitative assessment based on 2D photography performed by blinded panel 2. Physician – Global Aesthetic Improvement Scale Scores (P-GAIS) 3. Subject – Global Aesthetic Improvement Scale Scores (S-GAIS) 4. Physician – Global Satisfaction Questionnaire (P-GSQ) 5. Subject – Global Satisfaction Questionnaire (S-GSQ) Each individual endpoint will be based on study subject population response for each individual endpoint. |
| | Safety: Safety will be evaluated using the following measures: 1. Numerical Rating Scale (NRS), a 10-point pain scale 2. Self-reported and observed adverse events Fundamental Also of interact is the elasticity measurement at Days 00 and 180 |
| STUDY DESIGN | This study is a prospective, single-center, open-label study for the evaluation of the ThermiRF device in the treatment of submental skin laxity. |
| INTERIM | No annual reports for the FDA are anticipated prior to the end of data collection and database lock due to the short nature of this study. |
| | A single interim analysis is planned to support a manuscript and presentation. Final study results will not be made available until post database lock. |
| FINAL ANALYSES | All final planned analyses identified in this SAP will be completed after the last subject has completed their 6 month follow up. |





# 3 SEQUENCE OF PLANNED ANALYSES

#### 3.1 INTERIM ANALYSES

#### 3.1.1 ANNUAL REPORTS

As this study is expected to be completed within one year, no annual reports are anticipated at this time.

#### 3.1.2 OTHER INTERIM REPORTS

timing of the interim report is expected to occur prior to database lock and prior to the final analysis. An aggregate review of data to support a publication and/or presentation is anticipated at this time. The

## 3.2 FINAL ANALYSES AND REPORTING

necessary. Any results from these unplanned analyses will also be clearly identified as post-hoc analyses to ThermiGen, LLC following database lock. Any post-hoc, exploratory analyses completed to support subject has completed the Day 180 follow-up visit. Key statistics and study results will be made available planned study analyses, which were not identified in this SAP, will be documented and reported as All final, planned, analyses identified in the protocol and in this SAP will be performed only after the last

# 4 STUDY OBJECTIVES AND ENDPOINTS

#### 4.1 STUDY OBJECTIVES

### 4.1.1 Primary Objective/Endpoint

as determined by a quantitative assessment based on 3D photography. The primary endpoint is an improvement of at least 20 mm<sup>2</sup> in overall lift of the submental area at Day 90

## 4.1.2 SECONDARY OBJECTIVE/ENDPOINTS

Days 90 and 180 evaluated by the investigator and subject using the following subjective assessments: The secondary endpoint is overall aesthetic improvement of the submental area and jawline definition at

- Qualitative assessment based on 2D photography performed by blinded panel
- Physician Global Aesthetic Improvement Scale Scores (P-GAIS)
- Subject Global Aesthetic Improvement Scale Scores (S-GAIS)
- 4. Physician Global Satisfaction Questionnaire (P-GSQ)
- Subject Global Satisfaction Questionnaire (S-GSQ)
- Each individual endpoint will be based on study subject population response for each individual endpoint.

#### 4.1.3 SAFETY ENDPOINTS

Numerical Rating Scale (NRS) as a 10-point pain scale The safety endpoints will be self-reported and observed adverse events along with the reporting of the





#### 5 SAMPLE SIZE

The null and alternative hypotheses are:

$$H_0$$
:  $\pi \le 0.45$  (or 45%) vs.  $H_a$ :  $\pi > 0.45$ 

where  $\pi$  is the true proportion of subjects with at least 20 mm<sup>2</sup> lift. Under the assumptions that

- 1.  $\pi = 0.70$  (or 70%) for subjects not prematurely withdrawing from the study; and
- 2. The dropout rate is 12.5% and all dropouts will be considered as non-responders

a sample of size 70 enrolled subjects provides approximately 85% power to reject the null hypothesis in favor of the alternative at a one-sided  $\alpha$ =0.05

### 6 ANALYSIS POPULATIONS

## 6.1 INTENT TO TREAT POPULATION (ITT)

be performed using this population. The intent-to-treat (ITT) population for this study includes all subjects that signed the informed consent form, meet inclusion/exclusion criteria, and are enrolled in the study. The primary efficacy analysis will

### 6.2 Per-Protocol Population (PP)

excluded medication, and do not have a major protocol violation (see Attachment 1). The per-protocol population (PP) for this study will include all subjects who have completed the Day 90 visit, have an evaluable photograph to measure the area of lift from the Day 90 visit, have not used an

#### 6.3 SAFETY

The safety population of this study will include all enrolled subjects who received at least one treatment

from section 8.6.2 of the clinical protocol has been included here for reference (Table 1). For clarification purposes of the analysis populations described in sections 6.1 - 6.3, the following table

Table 1. Subject Status Classification

| Classification | Criteria |
|-------------------------|----------------------------------------------|
| Screen Failure | Signs the ICD but does not meet entry |
| | criteria or withdraws prior to Visit 2. |
| Enrolled | Signs the ICD and met all |
| | inclusion/exclusion criteria |
| Treated | Signs the ICD and successfully completes V2 |
| Discontinued/Withdrawal | Signed the ICD but does not successfully |
| | complete any visits |
| Completed | Signs the ICD and successfully completes all |
| | study visits |





### 6.4 RATER AGREEMENT POPULATION

reliability among two unblinded clinicians and three blinded clinicians. For more details, see section to those taken at baseline and days 90 and 180. These photos will be used to test inter and intra rater Thirty subjects, chosen in sequential order of enrollment, will have 2D photos taken at Day 60 in addition

# GENERAL ISSUES FOR STATISTICAL ANALYSIS

#### 7.1 ANALYSIS SOFTWARE

datasets, tables, listings, figures and analyses. (BBA) will be programmed using SAS® Software version 9.4 or later or R version 3.2.3 or later. BBA Standard Operating Procedures (SOPs) will be followed in the creation and validation of all analysis Analysis data sets, statistical analyses and associated output generated by Boston Biomedical Associates

# 7.2 DISPOSITION OF SUBJECTS AND WITHDRAWALS

subject non-compliance, adverse event/serious adverse event, other). and by reason for discontinuation (subject withdrew consent, subject terminated prematurely by sponsor, number and percent of ITT subjects who prematurely withdrew from the study will be presented overall percent of ITT subjects who completed each scheduled assessment will be presented in a table. The accountability completeness, screen failures will also be presented. The frequency and percent of subjects in each analysis population (percentages will be based on number of enrolled subjects). The number and All subjects who provide written informed consent will be accounted for, and for purposes of subject

A flow chart and listing will also summarize subject accountability.

# METHODS FOR WITHDRAWALS, MISSING DATA, AND OUTLIERS

observations most likely will occur. For the primary analysis on the primary efficacy endpoint, missing remaining efficacy endpoints and for safety endpoints, there will be no imputation of missing data prior to the primary efficacy endpoint will also be carried out only on subjects with available data. For all subject has a Day 60 image evaluation but is missing the Day 90 image evaluation, the Day 60 evaluation data will be imputed as a non-responder (i.e., imputed as "less than 20 mm2 lift"). In the case that a All reasonable efforts will be made to obtain complete data for all subjects; however, missing will be carried forward in the primary endpoint analysis. As a sensitivity analysis, the primary analysis on

Tables detailing missing data and analysis populations will be provided in the final report

#### 7.4 PROTOCOL VIOLATIONS

subject from the PP analysis population are identified in a study evaluability checklist and are included in subjects (overall and by site) with each violation type. Major protocol violations that may exclude a Protocol violations will be summarized in the CSR. This summary will include the number and percent of





# 7.5 MULTIPLE COMPARISONS AND MULTIPLICITY

statistical testing in support of labeling claims. No adjustments for multiple comparison will be made, as secondary endpoints will not undergo formal

### 7.6 ASSESSMENT OF HOMOGENEITY

homogeneity across sex, age groups, and condition types will be performed as outlined in Section 12 As this is a single-site study, no analysis will be performed for site homogeneity. Assessment of

# DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS

#### 8.1 Demographics

categorical variables, the summary will include number and percent of ITT subjects summary will include sample size, mean, median, standard deviation, minimum and maximum. For pressure (mmHg) for all ITT subjects will be summarized in a table. For continuous variables, the ethnicity, height (inches), weight (lbs), BMI, heart rate (bpm), as well as systolic and diastolic blood Age at screening (in years), sex (Male, Female), race (Not Done, White, Black or African American, American Indian/Alaskan Native, Asian, Native Hawaiian or Other Pacific Islander, Unknown, Other),

# 8.2 Prior and Concurrent Medications

A listing will be provided detailing subjects' medications, but no table is planned at this time

### 8.3 BASELINE MEDICAL HISTORY

percent of subjects who do not have any history of the condition, who currently have the condition, and The medical history of all ITT subjects will be summarized in a table. For each condition, the number and who have a resolved history of the condition will be presented

### 8.4 SCREENING PHYSICAL EXAM

body system, the number and percentage of ITT subjects considered normal and abnormal will be All subjects will undergo a physical examination for examination of various body systems. For each

### 9 Treatment Details

For the ITT population, descriptive statistics of number of incisions made, number of RF passes minimum and maximum. These will be presented for right-lateral, frontal, left-lateral, and total will be presented. Descriptive statistics consist of sample size, mean, median, standard deviation, maximum temperature reached, average temperature reached, surface temperature, and time per unit area





## 10 EFFECTIVENESS ANALYSES

The following analyses will be carried out on the ITT and PP populations.

## 10.1 PRIMARY EFFECTIVENESS VARIABLE

90. The following hypothesis will be tested: The primary endpoint is an evaluation of the proportion of subjects with greater than 20 mm<sup>2</sup> lift at Day

 $H_0$ :  $\pi \le 0.45$  (or 45%) Ha:  $\pi > 0.45$  (or 45%)

binomial proportion test will be performed at  $\alpha$ =0.05. For the ITT population, the analysis will be carried 90% confidence interval of the percentage based on the exact binomial distribution. A one-sided exact include the number and percentage of subjects with greater than 20 mm<sup>2</sup> lift at Day 90 and a two-sided where  $\pi$  is the proportion of subjects with greater than 20 mm<sup>2</sup> lift at Day 90. Statistical summaries will out twice as follows:

- Any subject with missing data at Day 60 and Day 90 will be treated as non-response to the primary endpoint analysis. missing the Day 90 image evaluation, the Day 60 evaluation will be carried forward in the photography (primary analysis). In the case that a subject has a Day 60 image evaluation but is
- 2 will be carried forward in the primary endpoint analysis. has a Day 60 image evaluation but is missing the Day 90 image evaluation, the Day 60 evaluation Any subject with missing data at Day 60 and Day 90 will be removed. In the case that a subject

## 10.2 SECONDARY EFFECTIVENESS VARIABLES

missing data for a given variable will be excluded from analysis on that variable There will be no imputation of missing data before analyses on the following variables. Subjects with

## 10.2.1 Validation of Rater's Assessment

agreement among raters will validate the method. are from which visit. The other three will remain blinded to the visit. All raters will be compared using at both baseline and Day 60. Two of the five will be unblinded and will have knowledge of which photos To assess the rater's assessment of improvement, a total of five clinicians will review the 2D photography Cohen's unweighted kappa statistic. Based on the Landis et al. scale, a substantial or almost perfect

subjects in each of the 5 categories and the two-sided Clopper-Pearson 95% CI of the percentages. A the ITT and PP populations at each visit. The summary will include the number and percentage of Physician will report P-GAIS on a scale of 1-5 at Days 60, 90 and 180. Tables will summarize this in both binomial test of proportions will be carried out for those scoring 3 or greater verse those scoring 2 and 10.2.2 Physician — Global Aesthetic Improvement Scale Scores (P-GAIS)





# 10.2.3 Subject – Global Aesthetic Improvement Scale Scores (S-GAIS)

scoring 2 and lower. and percentage of subjects in each of the 5 categories and the two-sided Clopper-Pearson 95% CI of the summarize this in both the ITT and PP populations at each visit. The summary will include the number percentages. A binomial test of proportions will be carried out for those scoring 3 or greater verse those As in section 10.2.2, subjects will report S-GAIS on a scale of 1-5 at Days 60, 90 and 180. Tables will

# 10.2.4 Physician — Global Satisfaction Questionnaire (P-GSQ)

responding "Likely" or "Very Likely" verse all others. or "Very Satisfied" verse all others. Further, likelihood of recommendation will be tested amongst those proportions will be carried out to compare those assessed with improvement versus no improvement the categories and the two-sided Clopper-Pearson 95% CI of the percentages. A binomial test of Physician will fill out the P-GSQ at Days 60, 90 and 180. Tables will summarize this in both the ITT and Additionally, a binomial test of proportions will test satisfaction, by testing those grouped as "Satisfied" PP populations at each visit. The summary will include the number and percentage of subjects in each of

# 10.2.5 Subject – Global Satisfaction Questionnaire (S-GSQ)

or "Very Satisfied" verse all others. Further, likelihood of recommendation will be tested amongst those Additionally, a binomial test of proportions will test satisfaction, by testing those grouped as "Satisfied" proportions will be carried out to compare those assessed with improvement versus no improvement. the categories and the two-sided Clopper-Pearson 95% CI of the percentages. A binomial test of PP populations at each visit. The summary will include the number and percentage of subjects in each of Subjects will fill out the S-GSQ at Days 60, 90 and 180. Tables will summarize this in both the ITT and responding "Likely" or "Very Likely" verse all others

# 10.2.6 Qualitative Assessment Based on 2D Photography

sided Clopper-Pearson 95% CI of the percentages. Additionally, a binomial test of proportions will test The summary will include the number and percentage of subjects in each of the categories and the twoby reader and the median of the three readers by subject in both the ITT and PP populations at each visit. between the photos using a five-point scale (1= "Much Improved", 2= "Minimally Improved", 3= "No compare photographs and provide a qualitative assessment of overall improvement in submental area Subjects will have 2D photographs taken at screening, Day 90 and Day 180. A blinded panel will improvement, by testing those grouped as "Much Improved" or "Minimally Improved" verse all others Change from Baseline", 4= "Minimally Worse", 5= "Much Worse"). Tables will summarize the ratings

# 10.3 EXPLORATORY EFFICACY VARIABLE - ELASTICITY

at each visit. The two-sided 95% confidence interval of the means will be presented. standard deviation, minimum, maximum) of elasticity and of the change from baseline will be presented Elasticity is collected at baseline and Days 90 and 180. Descriptive statistics (sample size, mean, median





#### 11 SAFETY ANALYSIS

be performed on the Safety Population. Activities (MedDRA) central coding dictionary, version 19.1 or greater. All analyses described below will All adverse events (AEs) will be coded using the standardized Medical Dictionary for Regulatory

## 11.1 NUMERICAL RATING SCALE (NRS)

summarized. The summary consists of the sample size, mean, median, standard deviation, minimum and NRS will be summarized for the Safety Population at Days 30, 60 (on the sample of size 30), 90, and 180 Change from Day 30 to Days 60, 90 and 180, and change from Day 90 to Day 180 will also be

#### 11.2 ALL ADVERSE EVENTS

provided will be the percent of subjects in the Safety Population experiencing one or more adverse events. provide both the number of subjects and the number of events within a reporting period. Percentages treatment emergent adverse event is defined as an event that started or worsened in severity at or after the emergent AEs (TEAE) by System Organ Class (SOC) and Preferred Term (PT) will be prepared. A Summaries of incidence rates and relationship to the investigational device of individual treatment first attempt at treatment. Because a subject may experience more than one TEAE, summaries will

SOC and PT, the severity of AE, whether or not the AE is classified as serious (SAE), the relationship of the AE to the investigational device or procedure, the action taken, the outcome, and the adjudication A listing of all adverse events will include the subject number, AE number, days since procedure, the AE

AEs will be recorded for all enrolled subjects to time of withdrawal, and reported in a table for all Safety

# 11.3 ADVERSE EVENTS LEADING TO WITHDRAWAL

also be provided, displaying details of the event(s) captured on the CRF SOC and PT will be prepared for the Safety Population. A data listing of AEs leading to withdrawal will A summary of incidence rates (frequencies and percentages) of TEAEs leading to study withdrawal, by

## 11.4 SERIOUS ADVERSE EVENTS (SAE)

subjects and the number of events within a reporting period. Percentages provided will be the percent of subjects experiencing one or more serious adverse events. A data listing of SAEs will also be provided, serious TEAEs SAEs by SOC and PT will be prepared. Summaries will provide both the number of Summaries of incidence rates and relationship to the investigational device/procedure of individual displaying details of the event(s) captured on the CRF.

# 11.5 DEVICE OR PROCEDURE RELATED ADVERSE EVENTS

reporting period. Percentages provided will be the percent of subjects experiencing one or more device or prepared. Summaries will provide both the number of subjects and the number of events within a Summaries of incidence rates of device and procedure related AEs and SAEs by SOC and PT will be





provided, displaying details of the event(s) captured on the CRF procedure related adverse events. Data listings of device and procedure related AEs and SAEs will also be

#### 11.6 Deaths

listing. Should any subjects die during the course of this study, relevant information will be supplied in a data

# 12 PLANNED SUBGROUP ANALYSES

#### 12.1 SEX

secondary efficacy endpoints will be evaluated for each sex separately with the results side by side and the subgroups of sex. presented in a table for the ITT analysis set. The purpose of this analysis is to assess consistency across To understand any potential sex differences which may be relevant to this study, the primary and

#### 12.2 AGE

analysis that creates an even dichotomous split) separately with the results side by side and presented in a primary and secondary efficacy endpoints will be evaluated for age groupings (to be determined at time of table for the ITT analysis set. The purpose of this analysis is to assess consistency across the subgroups of To understand any potential differences amongst age groups which may be relevant to this study, the

#### 12.3 Per-Protocol

populations. As stated in previous sections, all secondary endpoint analysis will be reported in both the ITT and PP

Additional subgroup or exploratory analyses may be completed following database lock

### 13 REPORTING CONVENTIONS

planned shells of output for the study report is provided in Attachment 2 All reporting will meet the standards of BBA SOP BS002 and its associated work instructions. The

## 13.1 OTHER REPORTING CONVENTIONS

- such that Landscape orientation would be easier to interpret. Tables, figures, and listings will be All tables, figures, and data listings will be presented in Portrait Orientation, unless dimensions are presented on a single page whenever possible.
- Each table will have a supporting data listing.
- Legends will be used for all figures with more than one variable or item displayed
- preferred for all dates. All date values will be presented as DDMMMYYYYY (e.g., 29AUG2001) format. A four-digit year is
- of each page of output. The analysis population will be identified at the top of all tables, figures, and All tables, figures, and data listings will have a version identifier and date/time stamp on the bottom
- The margins of all tables, figures, and listings will be 0.5-1 inch overall





- The text of tables and listings will be Times New Roman, 8-12 point.
- each category if >2 categories, of most important category if 2 categories. Unless otherwise specified in this SAP, all categorical variable summaries will include % (n/N) of
- standard deviation, N, median, minimum, and maximum. Unless otherwise specified in this SAP, all continuous variable summaries will include the mean,
- the CRF, while median, mean and standard deviation will be reported with have one more decimal Minimum and maximum will be reported with the number of significant figures as was reported on place than the data.
- Percentages will be reported to one decimal place, unless more precision is required for accuracy.
- values that are less than 0.001 will be reported as <0.001. P-values will be reported to three decimal places with a leading zero (for example, 0.032). Any p-





### ATTACHMENT 1. MAJOR PROTOCOL DEVIATIONS EVALUABILITY CHECKLIST

Attached to SAP as a reference.





# ATTACHMENT 2. TABLE, FIGURE, AND LISTING SHELLS

Attached to SAP as a reference.

#### Appendix 1: Evaluability Checklist for Definition of Deviations (Major vs. Minor)

| DEVIATION CATEGORY | DEVIATION<br>SUBCATEGORY | Selected for<br>study?<br>Yes/No | MEETS THE<br>DEFINITION OF<br>MAJOR? | EXCLUDED<br>FROM PER<br>PROTOCOL<br>ANALYSIS? |
|---|---|---|---|---|
| INFORMED CONSENT | | Yes | | |
| Dala Dasmansible for Identification and Treatings | a. Signed informed consent/assent not available on site | Yes | Y | Y |
| Role Responsible for Identification and Tracking: Sponsor Clinical | b. Wrong informed consent/assent version signed | Yes | Y | Y |
| Method of Identification: Direct review of each subject's signed ICF | c. Informed consent not signed and/or dated by subject (or parent/Legally Acceptable representative, if applicable) | Yes | Y | Y |
| | d. Informed consent/assent not signed and/or dated by appropriate site staff. | Yes | Y | N |
| | e. Informed consent/assent not signed prior or at Visit 1 following any study procedure | Yes | Y | Y |
| Study Specific Details and Detionals | f. Other informed consent/assent deviations | Yes | Y | |

#### **Study Specific Details and Rationale:**

- A. Site to contact subject for copy of ICF for files If subject not provided copy of ICF or copy not available, follow instructions for C.
- B. Assess follow-up and signing of correct version.
- C. Follow-up and document reason for oversight, inform IRB as required. Counsel site.
- D. Assess impact with study team.

| ELIGIBILITY CRITERIA NOT MET | NA | Yes | Yes |
|------------------------------|----|-----|-----|

| DEVIATION CATEGORY | DEVIATION<br>SUBCATEGORY | Selected for<br>study?<br>Yes/No | MEETS THE<br>DEFINITION OF<br>MAJOR? | EXCLUDED<br>FROM PER<br>PROTOCOL<br>ANALYSIS? |
|---|---|---|---|---|
| Role Responsible for Identification and Tracking: Sponsor Clinical Method of Identification: Direct review of each subject's source records when able. | All eligibility criteria | Yes | Y | N |
| Direct review of electronic data file (remote desk monitoring) | Select eligibility criteria not met | N | Y | Y |

Study Specific Details and Rationale:
All eligibility criteria deviations are to be reviewed for consideration of important status.

| NOT WITHDRAWN AFTER DEVELOPING<br>WITHDRAWAL CRITERIA | | Yes | | |
|---|---|---|---|---|
| Role Responsible for Identification and Tracking: | a. Not withdrawn from study | Yes | Y | Y |
| Sponsor Clinical | b. Not discontinued from study treatment | Yes | Y | NA |
| Method of Identification: During monitoring visits, review of data. | c. Other deviation of not being withdrawn after developing withdrawal criteria | Yes | Y | NA |

#### **Study Specific Details and Rationale:**

All protocol specified withdrawal criteria should be reviewed to determine the status of "important" and if documentation exists supporting the non-withdrawal of the subject as well as discussions between the investigator and the sponsor.

| EXCLUDED MEDICATION OR DEVICE | Yes |
|-------------------------------|-----|

| DEVIATION CATEGORY | DEVIATION<br>SUBCATEGORY | Selected for<br>study?<br>Yes/No | MEETS THE<br>DEFINITION OF<br>MAJOR? | EXCLUDED<br>FROM PER<br>PROTOCOL<br>ANALYSIS? |
|---|---|---|---|---|
| Role Responsible for Identification and Tracking: | Medication or dose of medication, excluded by the protocol, was administered | Yes | Y | N |
| Sponsor Clinical | b. Device, excluded by the protocol, was administered (Example: received another device treatment during study conduct) | Yes | Y | Y |

#### **Study Specific Details and Rationale:**

All medication deviations should be reviewed to determine if documentation exists supporting the non-withdrawal of the subject as well as discussions between the investigator and the sponsor.

| VISIT COMPLETION | | Yes | | |
|---|---|---|---|---|
| Role Responsible for Identification and Tracking: | a. Missed visit at critical data point | Yes | Y | Y |
| Sponsor Clinical Method of Identification: | b. Missed any visit other than critical data point | Yes | Y | N |
| Data review. | c. Out of window visit/phone contact | Yes | N | N |

#### **Study Specific Details and Rationale:**

A. Missed visits will be reviewed for importance as follows: is there a pattern of non-compliance, was the visit missed due to an AE/SAE, or because of safety management guidance. Multiple missed consecutive visits/phone contact will be assessed. Team will review these categories during reviews and determine importance.

| ASSESSMENT OR TIME POINT COMPLETION | | Yes | | |
|---|---|---|---|---|
| Role Responsible for Identification and/or Tracking: | a. Missed critical assessment (e.g., Photos for critical timepoint, questionnaires) | Yes | Y | Y |
| | b. Incomplete assessment | Yes | Y | N |
| | c. Assessment not properly performed | Yes | Y | N |

| DEVIATION CATEGORY | DEVIATION<br>SUBCATEGORY | Selected for<br>study?<br>Yes/No | MEETS THE<br>DEFINITION OF<br>MAJOR? | EXCLUDED<br>FROM PER<br>PROTOCOL<br>ANALYSIS? |
|---|---|---|---|---|
| Sponsor clinical team | d. Out of window assessment (optional) | Yes | N | N |
| | e. Out of Window efficacy assessment ( <i>optional</i> ) | Yes | Y | N |
| Method of Identification: | f. Out of Window safety assessment (optional) | Yes | Y | N |
| Data review | g. Out of Window treatment administration ( <i>optional</i> ) | N/A | Y | N |

#### **Study Specific Details and Rationale:** Part 1:

Overall, assessments will be reviewed to determine if there is a general pattern of non-compliance which may be determined by the team to be Important. Missed VS and physical exam may impact subject safety if changes in these assessments cannot be evaluated. AEs must be assessed to determine safety of IP. Missed efficacy evaluations (i.e., questionnaires) will impact the data analysis and integrity of the study.

| FAILURE TO REPORT SAFETY EVENTS PER PROTOCOL | | Yes | | |
|---|---|---|---|---|
| Role Responsible for Identification and Tracking: | a. SAE Occurred but was not reported. SAE warranted subject be discontinued but subject was not discontinued | Yes | Yes | N |
| Investigator, sponsor clinical team | b. AEs of special interest not reported or not properly qualified by the PI for causality | Yes | No | N |
| Method of Identification: Review of safety reports (spontaneous or voluntary | c. Pregnancy occured | Yes | Yes | N |
| reports) | d. Other: Define: RASH (specific eCRF page) | Yes | Yes | N |
| Study Specific Details and Rationale: | | | | |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 1 | |
|-----------------------------------------------|-------------|
| Analysis Populations | |
| | % (n/N) |
| All Enrolled | XX |
| Intention to Treat Population (ITT) | XX.X (X/XX) |
| Per Protocol Population (PPP) | XX.X (X/XX) |
| Safety Population (SAF) | XX.X (X/XX) |
| Note: Percentages are based on "All Enrolled" | • |

| Listing 1<br>Analysis Populations | | | | |
|---|---|---|---|---|
| Subject ID | Subject ID Enrolled ITT PP SAF | | | |
| XX-XXX | Yes/No | Yes/No | Yes/No | Yes/No |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

Version: Protocol Rev. A; SAP Rev. B

| | | Table | e 2 | |
|---|---|---|---|---|
| Subject Accountability | | | | |
| | ITT Population | | | |
| Eligible Missed Complete Early Exit | | | | |
| Visit N | | % (n/N) | % (n/N) | % (n/N) |
| Screening | XXX | | | |
| Procedure | XX | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Day 30 | XX | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Day 60 | XX | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Day 90 | XX | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Day 180 | XX | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |

Note: Percentages are based on the number of subjects in the ITT Population.

| Listing 2 Subject Accountability | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Screening<br>Date | Procedure<br>Date | 30 Day Visit | 60 Day Visit | 90 Day Visit | 180 Day<br>Visit | Study Exit | Exit Reason |
| XX-XXX | Date9. | Date9. | Date9. | Date9. | Date9. | Date9. | Date9. | |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

Figure 1. Subject Accountability Flowchart



Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 3 Subject Demographics and Baseline Characteristics ITT Population | |
|---|---|
| 111 1 opulution | N=XX |
| Age (years) | |
| Mean $\pm$ SD (N) | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) |
| Sex | 111111 (1111, 1111) |
| Male | XX.X (X/XX) |
| Female | XX.X (X/XX) |
| Race | ` |
| White | XX.X(X/XX) |
| Black or African American | XX.X(X/XX) |
| American Indian/Alaskan Native | XX.X (X/XX) |
| Asian | XX.X(X/XX) |
| Native Hawaiian or Other Pacific Islander | XX.X(X/XX) |
| Other [1] | XX.X (X/XX) |
| Unknown/Not done | XX.X (X/XX) |
| Ethnicity | |
| Hispanic | XX.X(X/XX) |
| Non Hispanic | XX.X(X/XX) |
| Height (inches) | |
| Mean $\pm$ SD (N) | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) |
| Weight (lbs) | |
| Mean $\pm$ SD (N) | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) |
| BMI | |
| Mean $\pm$ SD (N) | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) |
| Heart Rate (bpm) | |
| Mean $\pm SD(N)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) |
| Blood Pressure - Systolic (mmHg) | |
| Mean $\pm$ SD (N) | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) |
| Blood Pressure - Diastolic (mmHg) | |
| Mean $\pm$ SD (N) | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) |

<sup>[1]</sup> See supportive listing for specific details

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | Listing 3 Subject Demographics and Baseline Characteristics | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Age | Sex | Race | Ethnicity | Height (in.) | Weight (lb.) | BMI | Heart Rate<br>(BPM) | SBP | DBP |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 4 | |
|---|---|
| Medical History | |
| ITT Population | |
| • | % (n/N) |
| Aesthetic Procedures to the Lower Part of the Face and Neck | |
| Current condition | XX.X(X/XX) |
| Past, resolved | XX.X(X/XX) |
| No prior history | XX.X (X/XX) |
| Injury to the Head | |
| Current condition | XX.X(X/XX) |
| Past, resolved | XX.X(X/XX) |
| No prior history | XX.X (X/XX) |
| Severe Solar Elastosis | |
| Current condition | XX.X(X/XX) |
| Past, resolved | XX.X(X/XX) |
| No prior history | XX.X (X/XX) |
| Facial Wounds or Acute Infections in the Lower Part of the Face or Neck | |
| Current condition | XX.X(X/XX) |
| Past, resolved | XX.X(X/XX) |
| No prior history | XX.X (X/XX) |
| Immunodeficiency | |
| Current condition | XX.X (X/XX) |
| Past, resolved | XX.X (X/XX) |
| No prior history | XX.X (X/XX) |
| Injury Requiring Implants or Metal Stents | |
| Current condition | XX.X(X/XX) |
| Past, resolved | XX.X(X/XX) |
| No prior history | XX.X (X/XX) |
| Cancer | |
| Current condition | XX.X(X/XX) |
| Past, resolved | XX.X (X/XX) |
| No prior history | XX.X (X/XX) |
| Cardiovascular Disease | |
| Current condition | XX.X(X/XX) |
| Past, resolved | XX.X(X/XX) |
| No prior history | XX.X (X/XX) |
| Allergies | 3/3/ 3/ (3//3/**) |
| Current condition | XX.X (X/XX) |
| Past, resolved | XX.X(X/XX) |
| No prior history | XX.X (X/XX) |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Psychiatric Disorders | |
|-----------------------|-------------|
| Current condition | XX.X (X/XX) |
| Past, resolved | XX.X (X/XX) |
| No prior history | XX.X (X/XX) |
| Congenital Anomaly | |
| Current condition | XX.X (X/XX) |
| Past, resolved | XX.X (X/XX) |
| No prior history | XX.X (X/XX) |
| Other [2] | |
| Current condition | XX.X (X/XX) |
| Past, resolved | XX.X (X/XX) |
| No prior history | XX.X (X/XX) |

<sup>[1]</sup> Subjects may have multiple past conditions, but will only be accounted for once for each separate condition with "Current" superseding "Past, resolved".

<sup>[2]</sup> See supporting listing for details

| | Listing 4 Medical History | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID Aesthetic Procedures to the Lower Part of the Face and Neck Subject ID Neck Face and Neck | | | | | | | | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 5<br>Screening Physical Exam<br>ITT Population | |
|---|---|
| | % (n/N) |
| Eyes | |
| Normal | XX.X (X/XX) |
| Abnormal | XX.X (X/XX) |
| Not Done | XX.X (X/XX) |
| Ears, Nose, Throat | |
| Normal | XX.X (X/XX) |
| Abnormal | XX.X (X/XX) |
| Not Done | XX.X (X/XX) |
| Head and Neck | |
| Normal | XX.X (X/XX) |
| Abnormal | XX.X (X/XX) |
| Not Done | XX.X (X/XX) |
| Heart | |
| Normal | XX.X (X/XX) |
| Abnormal | XX.X (X/XX) |
| Not Done | XX.X (X/XX) |
| Chest and Lungs | |
| Normal | XX.X(X/XX) |
| Abnormal | XX.X (X/XX) |
| Not Done | XX.X (X/XX) |
| Abdomen | |
| Normal | XX.X (X/XX) |
| Abnormal | XX.X (X/XX) |
| Not Done | XX.X (X/XX) |
| General Appearance | |
| Normal | XX.X (X/XX) |
| Abnormal | XX.X (X/XX) |
| Not Done | XX.X (X/XX) |

| Listing 5<br>Screening Physical Exam | | | | | | | |
|---|---|---|---|---|---|---|---|
| Subject ID | Fars Nose Head and Chest and General | | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | | Table 6<br>Treatment Details<br>ITT Population | | |
|---|---|---|---|---|
| | Right-lateral (N=XX) | Frontal (N=XX) | Left-Lateral (N=XX) | Total (N=XX) |
| Number of Incisions | | | | |
| $Mean \pm SD(N)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) |
| Number of RF Passes | | | | |
| $Mean \pm SD(N)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) |
| Maximum Temperature Reach | ned | | | |
| $Mean \pm SD(N)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) |
| Average Temperature Reache | d | | | |
| $Mean \pm SD(N)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) |
| Surface Temperature | | | | |
| $Mean \pm SD (N)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) |
| Time per Unit Area | | | · | · |
| $Mean \pm SD(N)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) | XX.X (XX, XX) |

| | Listing 6a Treatment Details | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Right - Lateral Frontal | | | | | | | | Left-La | teral | | | | | | | | |
| Subject ID | Subject ID # # Avg. Max. Surface Incisions Passes Temp Temp Temp. Time Incisions Passes Temp Temp. Time Incisions Passes Temp Temp. | | | | #<br>Incisions | #<br>Passes | Avg.<br>Temp | Max.<br>Temp | Surface<br>Temp. | Time | | | | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

| Listing 6b Treatment Details | | | | | | |
|---|---|---|---|---|---|---|
| | Total | | | | | |
| Subject ID | Subject ID # Incisions # Passes Avg. Temp Max. Temp Surface Temp. Time | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 7.1<br>Study Endpoints - Primary Endpoint<br>ITT Population | | | | |
|---|---|---|---|---|
| Population One-sided p-value [1] Population | | | | |
| Improvement ≥ 20 mm² at Day 90 | ITT (missing subjects as failures) | XX.X (X/XX) | X.XXX | (X.X, X.X) |
| | Subjects with Day 90 missing data | XX | | |
| | Subjects with Day 60 data carried forward | XX | | |
| Improvement ≥ 20 mm² at Day 90 | ITT (excluding missing subjects) | XX.X (X/XX) | X.XXX | (X.X, X.X) |
| | Subjects with Day 60 data carried forward | XX | | |

<sup>[1]</sup> Null hypothesis is that the true percentage of subjects with  $\geq 20 \text{ mm}^2$  improvement is less than or equal to 45%.

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval of the percent of subjects with improvement.

| Listing 7.1 | | | | |
|---|---|---|---|---|
| | Study Endpoints - Primary Endpoint | | | |
| Subject ID | Subject ID Analysis Population Day 60 Improvement Day 90 Improvement Endpoint | | | |
| XX-XXX | XX | XX or N/A | XX or Missing | XX |

P-value is calculated based on the one-sided exact binomial test.

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 7.1.1 Study Endpoints – Qualitative Assessment for the 2D Imaging ITT Population [1] | | |
|---|---|---|
| | Percent Agreement | Kappa Statistic [2] |
| Overall | | |
| | XX.X (X/XX) | X.XXX |
| Subgroups [3] | | |
| Reader 1-2 | XX.X (X/XX) | X.XXX |
| Reader 1-3 | XX.X (X/XX) | X.XXX |
| Reader 1-4 | XX.X (X/XX) | X.XXX |
| Reader 1-5 | XX.X (X/XX) | X.XXX |
| Reader 2-3 | XX.X (X/XX) | X.XXX |
| Reader 2-4 | XX.X (X/XX) | X.XXX |
| Reader 2-5 | XX.X (X/XX) | X.XXX |
| Reader 3-4 | XX.X (X/XX) | X.XXX |
| Reader 3-5 | XX.X (X/XX) | X.XXX |
| Reader 4-5 | XX.X (X/XX) | X.XXX |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> Readers 1 and 2 were unblinded to image visit date, Readers 3, 4, and 5 were blinded to image visit date.

| Listing 7.1.1 Study Endpoints – Qualitative Assessment for the 2D Imaging | | | | | | |
|---|---|---|---|---|---|---|
| Subject ID | Subject ID Analysis Population Reader 1 Reader 2 Reader 3 Reader 4 Reader 5 | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX |

<sup>[2]</sup> Readers compared using Cohen's unweighted Kappa statistic

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 7.1.2 Study Endpoints – Qualitative Assessment for the 2D Imaging at Day 60 ITT Population [1] | | | | | |
|---|---|---|---|---|---|
| Reader 1 [2] Reader 2 [2] Reader 3 [3] Reader 4 [3] Reader 5 [3] | | | | | |
| Based on your perceived Baseline vs. Day 60, how would you rate observed submental area change at Day 60? | | | | | |
| Much Improved | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Minimally Improved | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X(X/XX) | XX.X(X/XX) |
| No change from Baseline | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X(X/XX) | XX.X(X/XX) |
| Minimally Worse | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Much Worse | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> Reader blinded to image visit date.

| Listing 7.1.2 | | | | | | |
|---|---|---|---|---|---|---|
| Study Endpoints – Qualitative Assessment for the 2D Imaging | | | | | | |
| Subject ID Analysis Population Reader 1 Reader 2 Reader 3 Reader 4 Reader 5 | | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX |

<sup>[2]</sup> Reader unblinded to image visit date.

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 7.2.1 Secondary Endpoint – P-GAIS ITT Population with Available Data | | | | | | |
|---|---|---|---|---|---|---|
| | Day 60 [1] Day 90 Day 180 | | | | | |
| Assessment | | 95% CI[2] | | 95% CI[2] | | 95% CI[2] |
| Physician - Global Aesthetic Improvement Scale (P-GAIS) | | | | | | |
| 5 (Very Much Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 4 (Much Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 3 (Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 2 (No Change) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 1 (Worse) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [3] | X.XXX | | X.XXX | | X.XXX | |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> p-value from Binomial Proportion Test for proportion of subjects who have at least "Improved" [score of 3 or greater]

| Listing 7.2.1 | | | | |
|---|---|---|---|---|
| Secondary Endpoint – P-GAIS | | | | |
| Subject ID | Subject ID Analysis Population Day 60 [1] Day 90 Day 180 | | | |
| XX-XXX | XX | XX | XX | XX |

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | | Study End | able 7.2.2<br>dpoints - S-GAIS<br>n with Available Data | | | |
|---|---|---|---|---|---|---|
| Day 60 [1] Day 90 Day 180 | | | | | | |
| Assessment | | 95% CI [2] | | 95% CI [2] | | 95% CI [2] |
| Subject - Global Aesthetic Improvement Scale (S-GAIS) | | | | | | |
| 5 (Very Much Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 4 (Much Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 3 (Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 2 (No Change) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 1 (Worse) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [3] | X.XXX | | X.XXX | | X.XXX | |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> p-value from Binomial Proportion Test for proportion of subjects who have at least "Improved" [score of 3 or greater]

| Listing 7.2.2 | | | |
|---|---|---|---|
| Secondary Endpoint – S-GAIS | | | |
| Subject ID Day 60 [1] Day 90 Day 180 | | | |
| XX-XXX | XX | XX | XX |

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.
Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | Study Enc<br>ITT Population | ble 7.2.3<br>lpoints - P-GSQ<br>with Available Da | ata | | | |
|---|---|---|---|---|---|---|
| | Day 60 | [1] | Day 90 | | Day 180 | |
| Assessment | | 95% CI [2] | | 95% CI [2] | | 95% CI [2] |
| Physician - Global Satisfaction Questionnaire (P-GSQ) | <u>'</u> | | | | | • |
| When looking at the photo images and respective to your clinician assess | sment during this visit, do yo | ou see any change o | n the treated area with resp | pect to "improveme | ent" of the skin and overa | ll area? |
| Yes, if "yes" please check all that apply: | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Less sagging on the jawline and cheeks | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Tighter/lift under the chin area | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Smoother skin texture | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Jaw line more defined | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Less wrinkles/lines | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Other | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [3] | X.XXX | X . | X.XXX | | X.XXX | • |
| Compared to "BEFORE" treatment how does the subject's skin feel to | day (check all that apply? | | | | | |
| Tighter | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Firmer | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Smoother | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| No change from prior to treatment | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| How satisfied are you with the results of the treatment? | | | | | | |
| Very Satisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Satisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Neutral | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Dissatisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Very Dissatisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [4] | X.XXX | ζ | X.XXX | | X.XXX | · |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

<sup>[3]</sup> p-value from Binomial Proportion Test for proportion of subjects who were marked "Improved"

<sup>[4]</sup> p-value from Binomial Proportion Test for proportion of subjects who were marked "Satisfied" or "Very Satisfied" and "Likely" or "Very Likely"

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | Listing 7.2.3 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Study Endpoints - P-GSQ | | | | | | | | | |
| | | | Da | y 60 [1] | Day 90 | | | Day 180 | | |
| Subject | Analysis | Improvement? | Skin | Satisfaction? | Improvement? | Skin | Satisfaction? | Improvement? | Skin | Satisfaction? |
| ID | Population | (All reasons) | Feel? | Satisfaction: | (All reasons) | Feel? | Satisfaction: | (All reasons) | Feel? | Satisfaction: |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | | ole 7.2.4<br>points - S-GSQ | | | | |
|---|---|---|---|---|---|---|
| | | with Available Dat | | | | |
| | Day 60 | [1] | Day 90 | ) | Day 18 | 0 |
| Assessment | | 95% CI [2] | | 95% CI [2] | | 95% CI [2] |
| Subject - Global Satisfaction Questionnaire (S-GSQ) | | | | | | |
| Have you noticed any change with respect to "improvement" of the | skin appearance of your neck? | | | | | |
| Yes, if "yes" please check all that apply: | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Less sagging on the jawline and cheeks | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Tighter/lift under the chin area | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Smoother skin texture | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Jaw line more defined | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Less wrinkles/lines | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Other | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [3] | X.XXX | X.XXX X.XXX | | | X.XXX | ζ |
| Compared to "BEFORE" treatment how does your skin feel today ( | check all that apply? | | | | | |
| Tighter | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Firmer | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Smoother | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Make-up application easier | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Shaving easier | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No change from prior to treatment | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| How satisfied are you with the results of your treatment? | • | | | | | |
| Very Satisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Satisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Neutral | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Dissatisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Very Dissatisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [4] | X.XXX | ζ. | X.XXX | ζ. | X.XXX | ζ. |
| How likely are you to recommend this treatment to family and frien | ds? | • | | | | |
| Very Likely | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Likely | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Neutral | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Unlikely | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Very Unlikely | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [4] | X.XXX | | X.XXX | | X.XXX | |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

<sup>[3]</sup> p-value from Binomial Proportion Test for proportion of subjects who were marked "Improved"

<sup>[4]</sup> p-value from Binomial Proportion Test for proportion of subjects who were marked "Satisfied" or "Very Satisfied" and "Likely" or "Very Likely"

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | Listing 7.2.4 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Endpoints - S-GSQ | | | | | | | | | | | | |
| | Day 60 [1] Day 90 | | | | | | D | ay 180 | | | | | |
| Subject<br>ID | Analysis<br>Population | Improvement?<br>(All reasons) | Skin<br>Feel? | Satisfaction? | Recommend? | Improvement?<br>(All reasons) | Skin<br>Feel? | Satisfaction? | Recommend? | Improvement?<br>(All reasons) | Skin<br>Feel? | Satisfaction? | Recommend? |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

**Protocol:** An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

| | | | Table 7.2.5 | | | | | |
|---|---|---|---|---|---|---|---|---|
| S4 | tudy Endpoints – Qualitat | tivo Assossment | Table 7.2.5 | ng at Day 00 an | d Day 190 sampa | nad ta Dasalina | | |
| 50 | ludy Endpoints – Quanta | iive Assessineiii | ITT Populatio | | ш Бау тоо сошра | reu to baseille | | |
| | | | 1111 Topulatio | | ıv 90 | | | |
| | Reader 1 | 95% CI [1] | Reader 2 | 95% CI [1] | Reader 3 | 95% CI [1] | Total [3] | 95% CI [1] |
| Much Improved | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Minimally Improved | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No change | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Minimally Worse | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Much Worse | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Improvement | | | | | | | | |
| Yes | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [2] | X.XXX | | X.XXX | | X.XXX | | X.XXX | |
| | | | | Da | y 180 | | | |
| Much Improved | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Minimally Improved | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No change | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Minimally Worse | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Much Worse | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Improvement | | | | | | | | |
| Yes | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [2] | X.XXX | | X.XXX | | X.XXX | | X.XXX | |

<sup>[3]</sup> Median of 3 Reader's scores

| Listing 7.2.5 Study Endpoints – Qualitative Assessment for the 2D Imaging | | | | | | | |
|---|---|---|---|---|---|---|---|
| | | Day 90 Day 180 | | | | | Day 90 |
| Subject ID | Analysis Population | Reader 1 | Reader 2 | Reader 3 | Reader 1 | Reader 2 | Reader 3 |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX |

<sup>[1]</sup> Two-sided 95% Clopper-Pearson confidence interval.
[2] p-value from Binomial Proportion Test for proportion of subjects who were marked "Much Improved" or "Minimally Improved"

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift


## Table 7.3 Study Endpoints - Exploratory Endpoint Elasticity ITT Population with Available Data

| | Baseline<br>N= | | Day 90<br>N= | | Day 180<br>N= | |
|---|---|---|---|---|---|---|
| Assessment | Mean ± SD (N)<br>Median (Min, Max) | 95% CI [1] | Mean ± SD (N)<br>Median (Min, Max) | 95% CI [1] | Mean ± SD (N)<br>Median (Min, Max) | 95% CI [1] |
| Elasticity | <u>'</u> | • | | | | • |
| R0 | $XX.X \pm XX.X (XX)$ $XX.X (XX, XX)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) | $XX.X \pm XX.X (XX)$ $XX.X (XX, XX)$ | (X.X, X.X) |
| R2 | $XX.X \pm XX.X (XX) XX.X (XX, XX)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |
| R5 | $XX.X \pm XX.X (XX)$ $XX.X (XX, XX)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |
| R7 | $XX.X \pm XX.X (XX) XX.X (XX, XX)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |
| R9 | $XX.X \pm XX.X (XX)$ $XX.X (XX, XX)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |
| <b>Change from Baseline Elasticity</b> | | | | | | |
| R0 | N/A | N/A | $XX.X \pm XX.X (XX)$ $XX.X (XX.X, XX.X)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |
| R2 | N/A | N/A | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |
| R5 | N/A | N/A | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |
| R7 | N/A | N/A | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |
| R9 | N/A | N/A | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX, XX) | (X.X, X.X) |

<sup>[1]</sup> Two-sided 95% confidence interval of the percentage or the mean.

| | Listing 7.3 | | | |
|---|---|---|---|---|
| Study Endpoints - Exploratory Endpoint Elasticity | | | | |
| Subject ID | Analysis Population | Baseline | Day 90 | Day 180 |
| Subject ID | Amarysis i opulation | Bascinic | (Change from Baseline) | (Change from Baseline) |
| XX-XXX | XX | XX | XX | XX |
| ΑΛ-ΑΛΛ | ΛΛ | AA | (XX) | (XX) |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

Figure 2. Bar chart for R0 and R9 output



Figure 3. Bar chart for R2, R5, and R7 output



Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 8.1.1 Study Endpoints by Sex - Primary Endpoint ITT Population | | | |
|---|---|---|---|
| | Population | Male<br>% (n/N)<br>95% CI [1] | Female<br>% (n/N)<br>95% CI [1] |
| Improvement ≥ 20 mm <sup>2</sup> at Day 90 | ITT (missing subjects as failures) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX<br>(X.X, X.X)) |
| | Subjects with missing data | XX | XX |
| | Subjects with Day 60 data carried forward | XX | XX |
| Improvement ≥ 20 mm <sup>2</sup> at Day 90 | ITT (excluding missing subjects) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) |
| | Subjects with Day 60 data carried forward | XX | XX |

<sup>[1]</sup> Two-sided 95% Clopper-Pearson confidence interval.

| | Listing 8.1.1 | | | | |
|---|---|---|---|---|---|
| | Study Endpoints by Sex - Primary Endpoint | | | | |
| Subject ID | Sex | Analysis Population | Day 60 Improvement [1] | Day 90 Improvement | Endpoint |
| XX-XXX | XX | XX | XX or N/A | XX or Missing | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift


| | | <b>Table 8.2.1.1</b> | | | | |
|---|---|---|---|---|---|---|
| | Study En | dpoints by Sex - P- | GAIS | | | |
| | ITT Popul | ation with Availabl | le Data | | | |
| Day 60 [1] Day 90 Day 180 | | | | | | |
| | Male | Female | Male | Female | Male | Female |
| Assessment | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] |
| Physician - Global Aesthetic Improvement Scale ( | | | | | | |
| 5 (Very Much Improved) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) |
| 4 (Much Improved) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) |
| 3 (Improved) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) |
| 2 (No Change) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) |
| 1 (Worse) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

| | Listing 8.2.1.1 | | | | |
|---|---|---|---|---|---|
| | Secondary Endpoint by Sex – P-GAIS | | | | |
| Subject ID | Sex | <b>Analysis Population</b> | Day 60 [1] | Day 90 | Day 180 |
| XX-XXX | XX | XX | XX | XX | XX |

(X.X, X.X)

(X.X, X.X)

(X.X, X.X)

(X.X, X.X)

(X.X, X.X)

(X.X, X.X)

**Protocol:** An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental


| | | <b>Table 8.2.1.2</b> | | | | |
|---|---|---|---|---|---|---|
| | Study Endpoints by Sex – S-GAIS | | | | | |
| ITT Population with Available Data | | | | | | |
| Day 60 [1] Day 90 Day 180 | | | | | | |
| Male Female Male Female Male Female | | | | | | |
| Assessment | % (n/N) | % (n/N) | % (n/N) | % (n/N) | % (n/N) | % (n/N) |
| | 95% CI [2] | 95% CI [2] | 95% CI [2] | 95% CI [2] | 95% CI [2] | 95% CI [2] |
| Subject - Global Aesthetic Improvement Scale (S-GAIS) | | | | | | |
| 5 (Very Much Improved) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| 4 (Much Improved) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| 3 (Improved) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| 2 (No Change) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| 1 (Worse) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

| | Listing 8.2.1.2 | | | | |
|---|---|---|---|---|---|
| | Secondary Endpoint by Sex – S-GAIS | | | | |
| Subject ID | Subject ID Sex Analysis Population Day 60 [1] Day 90 Day 180 | | | | |
| XX-XXX | XX | XX | XX | XX | XX |

**Protocol:** An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

| | G. | Table 8.2.1.3 | D 000 | | | |
|---|---|---|---|---|---|---|
| | | udy Endpoints by Sex<br>Population with Ava | | | | |
| | Day | 1 | | y 90 | Day | 180 |
| | Male | Female | Male | Female | Male | Female |
| Assessment | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] | % (n/N)<br>95% CI [2] |
| Physician - Global Satisfaction Questionnaire (P-C | | | | | | |
| When looking at the photo images and respective to y | | | | | | |
| Yes, if "yes" please check all that apply: | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| 70 7 1 117 | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Less sagging on the jawline and cheeks | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Tighter/lift under the chin area | XX.X (X/XX) | XX.X (X/XX) | XX.X(X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| righter/fift under the chin area | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Smoother skin texture | XX.X (X/XX) | XX.X (X/XX) | XX.X(X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Smoother skin texture | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| 1 6 1 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Jaw line more defined | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Less wrinkles/lines | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Other | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| No | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Compared to "BEFORE" treatment how does the su | | all that apply? | | | | |
| | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Tighter | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Firmer | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Smoother | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| No change from prior to treatment | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| How satisfied are you with the results of the treatmen | t? | | | | | |
| Very Satisfied | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| very Saustieu | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| 0 4 6 1 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Satisfied | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| N 4 1 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Neutral | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| D: 2.5.1 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Dissatisfied | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| ** *** | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Very Dissatisfied | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit. [2] Two-sided 95% Clopper-Pearson confidence interval.

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | Listing 8.2.1.3 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Study Endpoints - P-GSQ | | | | | | | | | |
| | Day 60 [1] Day 90 Day 180 | | | | | | | | | |
| Subject | Sex | Improvement? | Skin | Satisfaction? | Improvement? | Skin | Satisfaction 2 | Improvement? | Skin | Satisfaction? |
| ID | Sex | (All reasons) | All reasons) Feel? Satisfaction? Timprovement: Skill Satisfaction? S | | | | | | | |
| XX-XXX | XX | | | | | | | | | |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | | Table 9 2 1 4 | | | | |
|---|---|---|---|---|---|---|
| | Study F | Table 8.2.1.4<br>ndpoints by Sex – S-0 | 260 | | | |
| | | napoints by Sex – S-C<br>llation with Available | | | | |
| | | 60 [1] | | v 90 | Day | 190 |
| | Male | Female | Male | Female | Male | Female |
| Assessment | % (n/N) | % (n/N) | % (n/N) | % (n/N) | % (n/N) | % (n/N) |
| | 95% CI [2] | 95% CI [2] | 95% CI [2] | 95% CI [2] | 95% CI [2] | 95% CI [2] |
| Subject - Global Satisfaction Questionnaire (S-GSQ) | | | | | | |
| Have you noticed any change with respect to "improvement" of the sk | in appearance of your | neck? | | | | |
| | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Yes, if "yes" please check all that apply: | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Y 1 4 1 1 1 1 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Less sagging on the jawline and cheeks | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Tinkton /life don the chin and | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Tighter/lift under the chin area | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Smoother skin texture | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Silloother skill texture | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Jaw line more defined | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| jaw iiile iiioi e delilled | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Less wrinkles/lines | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Ecss withkies/filles | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Other | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Other | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| No | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Compared to "BEFORE" treatment how does your skin feel today (ch | | 1 | | 1 | 1 | 1 |
| Tighter | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| 1.8 | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Firmer | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Smoother | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Make-up application easier | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Shaving easier | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| No change from prior to treatment | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| 11 | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| How satisfied are you with the results of your treatment? | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Very Satisfied | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X) $XX.X (X/XX)$ | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) |
| Satisfied | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) | (A.A, A.A)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) | (A.A, A.A)<br>XX.X (X/XX) |
| Neutral | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | XX.X (X/XX) | (X,X,X,X)<br>XX.X(X/XX) | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) | (X.X, X.X)<br>XX.X (X/XX) |
| Dissatisfied | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| I | $(\Delta,\Delta,\Delta,\Delta)$ | $(\Lambda,\Lambda,\Lambda,\Lambda)$ | (A.A, A.A) | $(\alpha, \alpha, \alpha, \alpha)$ | $(\Delta,\Delta,\Delta,\Delta)$ | (23.23, 23.23) |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 8.2.1.4 Study Endpoints by Sex – S-GSQ ITT Population with Available Data | | | | | | |
|---|---|---|---|---|---|---|
| Day 60 [1] Day 90 Day 180 | | | | | | |
| | Male | Female | Male | Female | Male | Female |
| Very Dissatisfied | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Very Dissaustieu | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| How likely are you to recommend this treatment to family and friends? | | | | | | |
| V 1 :11 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Very Likely | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| T. Harlan | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Likely | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Nt1 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Neutral | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| 77 17 1 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Unlikely | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| X7 | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Very Unlikely | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

| | Listing 8.2.1.4 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Endpoints by Sex - S-GSQ | | | | | | | | | | | | |
| | Day 60 [1] Day 90 | | | | | | | D | ay 180 | | | | |
| Subject<br>ID | ' Nov 1 Natistaction? Recommend? 1 Natistaction? Recommend? | | | | | Recommend? | Improvement?<br>(All reasons) | Skin<br>Feel? | Satisfaction? | Recommend? | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

Table 8.2.1.5

Study Endpoints by Sex – Qualitative Assessment for the 2D Imaging at Day 90 and Day 180 compared to Baseline
ITT Population with Available Data

| | Read | der 1 | Rea | der 2 | Rea | nder 3 | Tota | al [3] |
|---|---|---|---|---|---|---|---|---|
| | Male | Female | Male | Female | Male | Female | Male | Female |
| Assessment | % (n/N) | % (n/N) | % (n/N) | % (n/N) | % (n/N) | % (n/N) | % (n/N) | % (n/N) |
| | 95% CI [1] | 95% CI [1] | 95% CI [1] | 95% CI [1] | 95% CI [1] | 95% CI [1] | 95% CI [1] | 95% CI [1] |
| | | | | Da | y 90 | | | |
| Much Improved | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Minimally Improved | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | (X.X, X.X)<br>XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | (X.X, X.X)<br>XX.X (X/XX)<br>(X.X, X.X) | (X.X, X.X)<br>XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) | XX.X (X/XX)<br>(X.X, X.X) |
| No change | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Minimally Worse | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Much Worse | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| | | | | Day | y 180 | | | |
| Much Improved | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Minimally Improved | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| No change | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Minimally Worse | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |
| Much Worse | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) | (X.X, X.X) |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> Median of 3 Readers Scores

| Listing 8.2.1.5 Study Endpoints by Sex – Qualitative Assessment for the 2D Imaging | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Day 90 Day 180 | | | | | |
| Subject ID | Sex | Analysis Population | Reader 1 | Reader 2 | Reader 3 | Reader 1 | Reader 2 | Reader 3 |
| XX-XXX | | | | | | | | |

<sup>[1]</sup> Two-sided 95% Clopper-Pearson confidence interval.

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift


| | Table 8.3.1 Study Endpoints by Sex - Exploratory Endpoint Elasticity ITT Population with Available Data | | | | | |
|---|---|---|---|---|---|---|
| | Base | eline | Day | y <b>90</b> | Day | 180 |
| | Male | Female | Male | Female | Male | Female |
| Assessment | | | | | | |
| Elasticity – by each paramet | ter | | L | | | |
| Mean ± SD (N)<br>Median (Min, Max) | $\begin{array}{c} XX.X \pm XX.X (XX) \\ XX.X (XX.X, XX.X) \end{array}$ | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) |
| 95% CI [1] | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| Change from Baseline Elas | ticity – by each parameter | , | | | | |
| Mean $\pm$ SD (N) Median (Min, Max) $N/A$ $N/A$ $N/A$ $N/A$ $XX.X \pm XX.X (XX)$ $XX.X \pm X$ | | | | | | |
| 95% CI [1] | N/A | N/A | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |

<sup>[1]</sup> Two-sided 95% confidence interval of the percentage or the mean.

| | | | Listing 8.3.1 | | |
|---|---|---|---|---|---|
| | Study Endpoints by Sex - Exploratory Endpoint Elasticity | | | | |
| Subject ID Sex Analysis Population Baseline Day 90 Day 180 | | | | | |
| Subject ID | SCA | Analysis I opulation | Dascille | (Change from Baseline) | (Change from Baseline) |
| XX-XXX | XX-XXX XX XX XX XX XX | | | | |
| ΛΛ-ΛΛΛ | AA | ΛΛ | ΛΛ | (XX) | (XX) |

NOTE: Tables 8.1.1, 8.2.1.1, 8.2.1.2, 8.2.1.3, 8.2.1.4 and 8.3.1 will be repeated for the Age (dichotomous or categorical group comparison) as 8.1.2, 8.2.2.1, 8.2.2.2, 8.2.2.3, 8.2.2.4, and 8.3.2 to support the planned subgroup analyses

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift


| Table 9.1 | | | | |
|---|---|---|---|---|
| Study Endpoints - Primary Endpoint PP Population | | | | |
| Population % (n/N) One-sided p-value[1] 95% CI[2] | | | | |
| Improvement ≥ 20 mm2 at Day 90 | PP | XX.X (X/XX) | X.XXX | (X.X, X.X) |

<sup>[1]</sup>Null hypothesis is that the true percentage of subjects with ≥ 20 mm2 improvement is less than or equal to 45%.

P-value is calculated based on the one-sided exact binomial test.

[2[ Two-sided 95% Clopper-Pearson confidence interval.

| | Listing 9.1 | | |
|---|---|---|---|
| | Study Endpoints - Primary Endpoint | | |
| Subject ID | Analysis Population | Day 90 Improvement | Endpoint |
| XX-XXX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 9.1.1 Study Endpoints – Qualitative Assessment for the 2D Imaging PP Population [1] | | |
|---|---|---|
| | Percent Agreement | Kappa Statistic [2] |
| Overall | | |
| | XX.X (X/XX) | X.XXX |
| Subgroups [3] | | |
| Reader 1-2 | XX.X (X/XX) | X.XXX |
| Reader 1-3 | XX.X (X/XX) | X.XXX |
| Reader 1-4 | XX.X (X/XX) | X.XXX |
| Reader 1-5 | XX.X (X/XX) | X.XXX |
| Reader 2-3 | XX.X (X/XX) | X.XXX |
| Reader 2-4 | XX.X (X/XX) | X.XXX |
| Reader 2-5 | XX.X (X/XX) | X.XXX |
| Reader 3-4 | XX.X (X/XX) | X.XXX |
| Reader 3-5 | XX.X (X/XX) | X.XXX |
| Reader 4-5 | XX.X (X/XX) | X.XXX |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> Readers 1 and 2 were unblinded to image visit date, Readers 3, 4, and 5 were blinded to image visit date.

| | Listing 9.1.1 Study Endpoints – Qualitative Assessment for the 2D Imaging | | | | | |
|---|---|---|---|---|---|---|
| Subject ID | Subject ID Analysis Population Reader 1 Reader 2 Reader 3 Reader 4 Reader 5 | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX |

<sup>[2]</sup> Readers compared using Cohen's unweighted Kappa statistic

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 9.1.2 Study Endpoints – Qualitative Assessment for the 2D Imaging PP Population [1] | | | | | |
|---|---|---|---|---|---|
| Reader 1 [2] | | | | | |
| Based on your perceived Baseline vs. Day 60, 1 | now would you rate ob | served submental a | area change at Day | 60? | |
| Much Improved | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| Minimally Improved | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) | XX.X (X/XX) |
| No change from Baseline $XX.X.(X/XX) = XX.X.(X/XX) = XX.X$ | | | | | |
| Minimally Worse | | | | | |
| Much Worse | | | | | |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

| | Listing 9.1,2 Study Endpoints – Qualitative Assessment for the 2D Imaging | | | | | |
|---|---|---|---|---|---|---|
| Subject ID | Subject ID Analysis Population Reader 1 Reader 2 Reader 3 Reader 4 Reader 5 | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX |

<sup>[2]</sup> Reader unblinded to image visit date.

<sup>[3]</sup> Reader blinded to image visit date.

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | | Secondary E | ble 9.2.1<br>ndpoint – P-GAIS<br>with Available Data | ı | | |
|---|---|---|---|---|---|---|
| Day 60 [1] Day 90 Day 180 | | | | | | |
| Assessment | | 95% CI[2] | | 95% CI[2] | | 95% CI[2] |
| Physician - Global Aesthetic I | mprovement Scale (P-GA | AIS) | | | | 1 |
| 5 (Very Much Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 4 (Much Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 3 (Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 2 (No Change) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 1 (Worse) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [3] | X.XX | XX | X. | XXX | X.XX | X |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> p-value from Binomial Proportion Test for proportion of subjects who have at least "Improved" [score of 3 or greater]

| | Listing 9.2.1 |
|---|---|
| | Secondary Endpoint – P-GAIS |
| Subject ID | Subject ID Analysis Population Day 60 [1] Day 90 Day 180 |
| XX-XXX | VV VVV VV VV VV |

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | | Study End | able 9.2.2<br>dpoints - S-GAIS<br>n with Available Data | | | |
|---|---|---|---|---|---|---|
| Day 60 [1] Day 90 Day 180 | | | | | | |
| Assessment | | 95% CI [2] | | 95% CI [2] | | 95% CI [2] |
| Subject - Global Aesthetic Im | provement Scale (S-GAI | (S) | | | | |
| 5 (Very Much Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 4 (Much Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 3 (Improved) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 2 (No Change) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| 1 (Worse) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [3] | X.XXX | | X.XXX | ζ. | X.XX | X |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> p-value from Binomial Proportion Test for proportion of subjects who have at least "Improved" [score of 3 or greater]

| | Listing 9.2.2 | | |
|---|---|---|---|
| Secondary Endpoint – S-GAIS | | | |
| Subject ID | Subject ID Day 60 [1] Day 90 Day 180 | | |
| XX-XXX | XX | XX | XX |

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental **Protocol:** 

| | Study End<br>PP Population | ble 9.2.3<br>points - P-GSQ<br>with Available Da | | | | |
|---|---|---|---|---|---|---|
| | Day 60 [ | 1] | Day 90 | | Day 180 | ) |
| Assessment | | 95% CI [2] | | 95% CI [2] | | 95% CI [2] |
| Physician - Global Satisfaction Questionnaire (P-GSQ) | 1 | | | | | • |
| When looking at the photo images and respective to your clinician assessment | nent during this visit, do yo | u see any change o | n the treated area with resp | ect to "improveme | ent" of the skin and overal | l area? |
| Yes, if "yes" please check all that apply: | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Less sagging on the jawline and cheeks | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Tighter/lift under the chin area | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Smoother skin texture | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Jaw line more defined | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Less wrinkles/lines | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Other | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [3] | X.XXX | | X.XXX | | X.XXX | |
| Compared to "BEFORE" treatment how does the subject's skin feel today | y (check all that apply? | | | | | |
| Tighter | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Firmer | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| Smoother | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X(X/XX) | (X.X, X.X) |
| No change from prior to treatment | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| How satisfied are you with the results of the treatment? | | | | | | |
| Very Satisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Satisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Neutral | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Dissatisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Very Dissatisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [4] | X.XXX | | X.XXX | | X.XXX | |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[3]</sup> p-value from Binomial Proportion Test for proportion of subjects who were marked "Improved"
[4] p-value from Binomial Proportion Test for proportion of subjects who were marked "Satisfied" or "Very Satisfied" and "Likely" or "Very Likely"

| | Listing 9.2.3 Study Endpoints - P-GSQ | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Day 60 [1] Day 90 Day 180 | | | | | | | ay 180 | | | |
| Subject | Analysis | Improvement? | Skin | Satisfaction? | Improvement? | Skin | Satisfaction? | Improvement? | Skin | Satisfaction? |
| ID | Population | (All reasons) | Feel? | Satisfaction: | (All reasons) | Feel? | Satisfaction: | (All reasons) | Feel? | Satisfaction: |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | Study End | ole 9.2.4<br>points - S-GSQ<br>with Available Data | 1 | | | |
|---|---|---|---|---|---|---|
| | Day 60 | [1] | Day 90 | ) | Day 180 | |
| Assessment | | 95% CI [2] | | 95% CI [2] | | 95% CI [2] |
| Subject - Global Satisfaction Questionnaire (S-GSQ) | | | | | | |
| Have you noticed any change with respect to "improvement" of the skin ap | pearance of your neck? | | | | | |
| Yes, if "yes" please check all that apply: | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Less sagging on the jawline and cheeks | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Tighter/lift under the chin area | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Smoother skin texture | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Jaw line more defined | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Less wrinkles/lines | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Other | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [3] | X.XXX | X.XXX | | X.XXX | | X |
| Compared to "BEFORE" treatment how does your skin feel today (check a | ll that apply? | | | | | |
| Tighter | XX.X (X/XX) | (X.X, X.X) | XX,X (X/XX) | (X.X, X.X) | XX,X (X/XX) | (X,X, X,X) |
| Firmer | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Smoother | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Make-up application easier | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Shaving easier | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No change from prior to treatment | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| How satisfied are you with the results of your treatment? | | | | | | |
| Very Satisfied | XX.X (X/XX) | (X.X, X.X) | XX,X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Satisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Neutral | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Dissatisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Very Dissatisfied | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [4] | X.XXX | X | X.XXX | ζ ΄ | X.XX | X |
| How likely are you to recommend this treatment to family and friends? | | | · | | <u> </u> | |
| Very Likely | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Likely | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Neutral | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Unlikely | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Very Unlikely | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [4] | X.XXX | | X.XXX | | X,XXX | |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

<sup>[2]</sup> Two-sided 95% Clopper-Pearson confidence interval.

<sup>[3]</sup> p-value from Binomial Proportion Test for proportion of subjects who were marked "Improved"

<sup>[4]</sup> p-value from Binomial Proportion Test for proportion of subjects who were marked "Satisfied" or "Very Satisfied" and "Likely" or "Very Likely"

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | Listing 9.2.4 | | |
|---|---|---|---|
| | Study Endpoints - S-GSQ | | |
| Day 60 [1] Day 90 Day 180 | | | |
| Subject<br>ID | Analysis<br>Population | Improvement? Skin Improvement? Skin Improvement? Skin | Recommend? |
| XX-XXX | | | |

**Protocol:** An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

| | Table 9.2.5 Study Endpoints – Qualitative Assessment for the 2D Imaging at Day 90 and Day 180 PP Population | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Day 90 | | | | | | |
| | Reader 1 | 95% CI [1] | Reader 2 | 95% CI [1] | Reader 3 | 95% CI [1] | Total [3] | 95% CI [1] |
| Much Improved | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Minimally Improved | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No change | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Minimally Worse | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Much Worse $\left( \begin{array}{c ccc} XX.X \left( X/XX \right) & (X.X,X.X) \\ \end{array} \right) \left( \begin{array}{c ccc} $ | | | | | | | | |
| Improvement | | | | | | | | |
| Yes | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [2] | X.XXX | | X.XXX | | X.XXX | | X.XXX | |
| | | | Day | 180 | | | | |
| Much Improved | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Minimally Improved | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No change | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Minimally Worse | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Much Worse | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| Improvement | | | | | | | | |
| Yes | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| No | No XX.X (X/XX) (X. | | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) | XX.X (X/XX) | (X.X, X.X) |
| p-value [2] | X.XXX | | | | | | | |

<sup>[3]</sup> Median of 3 Readers scores

| Listing 9.2.5 Study Endpoints – Qualitative Assessment for the 2D Imaging | | |
|---|---|---|
| | | Day 90 Day 180 |
| Subject ID | Analysis Population | |
| XX-XXX | XX | XX XX XX XX XX XX |

<sup>[1]</sup> Two-sided 95% Clopper-Pearson confidence interval.
[2] p-value from Binomial Proportion Test for proportion of subjects who were marked "Much Improved" or "Minimally Improved"

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | | | ble 9.3 | | | |
|---|---|---|---|---|---|---|
| | Study E | | oratory Endpoint Elastici<br>opulation | ty | | |
| | Baseline<br>N= | Baseline<br>N= | | | Day 180<br>N= | |
| Assessment | Mean ± SD (N)<br>Median (Min, Max) | 95% CI of<br>the Mean | Mean ± SD (N)<br>Median (Min, Max) | 95% CI of<br>the Mean | Mean ± SD (N)<br>Median (Min, Max) | 95% CI of<br>the Mean |
| Elasticity | (************************************** | | (,, | | (,, | , ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |
| R0 | $XX.X \pm XX.X (XX) XX.X (XX.X, XX.X)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$ $XX.X (XX.X, XX.X)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| R2 | $XX.X \pm XX.X (XX)$ $XX.X (XX.X, XX.X)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| R5 | $XX.X \pm XX.X (XX)$ $XX.X (XX.X, XX.X)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| R7 | $XX.X \pm XX.X (XX)$ $XX.X (XX.X, XX.X)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| R9 | $XX.X \pm XX.X (XX)$ $XX.X (XX.X, XX.X)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| Change from Baseline F | Elasticity | | | | | |
| R0 | N/A | N/A | $\begin{array}{c} XX.X \pm XX.X (XX) \\ XX.X (XX.X, XX.X) \end{array}$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| R2 | N/A | N/A | $XX.X \pm XX.X (XX)$ $XX.X (XX.X, XX.X)$ | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| R5 | N/A | N/A | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| R7 | N/A | N/A | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |
| R9 | N/A | N/A | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) | $XX.X \pm XX.X (XX)$<br>XX.X (XX.X, XX.X) | (X.X, X.X) |

<sup>[1]</sup> Two-sided 95% confidence interval of the percentage or the mean.

| | Listing 9.3 | | | |
|---|---|---|---|---|
| | Study Endpoints - Exploratory Endpoint Elasticity | | | |
| Subject ID | Subject ID Analysis Population Baseline Day 90 Day 180 (Change from Baseline) (Change from Baseline) | | | |
| XX-XXX | XX | XX | XX<br>(XX) | XX<br>(XX) |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

Figure 4. Bar chart for R0 and R9 output [PP Population]



Figure 5. Bar chart for R2, R5, and R7 output [PP Population]



Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| | Table 10 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Overall Treatment Emergent Adverse Events Summary [1] [2] | | | | | | | | | |
| Safety Population After Treatment After Day 30, After Day 60, After Day 90, Total | | | | | | | | | | |
| | After Treatment Prior to Day 30 Prior to Day 30 Prior to Day 60 Prior to Day 6 | | | | | | | | | |
| | N=XXX N=XXX N=XXX N=XXX | | | | | | | | | |
| | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | " w/Event | | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) |
| All Adverse Events | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| Device Related | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| Serious Adverse Events | Adverse Events XX XX.X (X/XX) XX | | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | |
| Device Related | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |

<sup>[1]</sup> Events reported as adjudicated or by site if not adjudicated

| | | I | Listing 10 | | | |
|---|---|---|---|---|---|---|
| | Summary of Adverse Events | | | | | |
| Subject ID | Adverse Event<br>Number | SOC<br>(Preferred Term) | Days Post<br>Procedure | Any Adverse<br>Event | Any Serious<br>Adverse<br>Event | Event Related to Study Treatment |
| XX-XXX | XXX XX XX XX XX XX | | | | | |

<sup>[2]</sup> Denominators of time points are subjects past the visit window or with an event

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift


| Overal | ll Treatment E | Emergent Adve | | Table 11<br>Summary by<br>Safety Populat | ion | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Prior | After Treatment Prior to Day 30 N=XX | | After Day 30,<br>up to Day 60<br>N=XX | | After Day 60,<br>up to Day 90<br>N=XX | | After Day 90,<br>up to day 180<br>N=XX | | Total<br>N=XX |
| | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) |
| All Adverse Events | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| SOC 1 | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| PT 1.1 | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| PT 1.2 | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| SOC 2 | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| PT 2.1 | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| PT 2.2 | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each System Organ Class | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each Preferred Term | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |

<sup>[1]</sup> Events reported as adjudicated or by site if not adjudicated

## NOTE: This SOC and PT structure to be carried forward to tables

| | | I | Listing 11 | | | |
|---|---|---|---|---|---|---|
| | Summary of Adverse Events by SOC and PT | | | | | |
| Subject ID Adverse Event Number Number SOC Days Post Procedure Event Procedure Procedure Event Event Event Event Event Event Related to Social Structure | | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX |

<sup>[2]</sup> Denominators of time points are subjects past the visit window or with an event

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Overall Tre | atment Emerge | ent Serious Ad | verse Eve | Table 12 | by System | Organ Class a | nd Prefer | red Term [1] [ | 21 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Safety Population | | | | | | | | | | |
| After Treatment Prior to Day 30 Up to Day 60 After Day 60, Up to Day 90 Up to day 180 Total up to day 180 | | | | | | | | | | |
| | 1 | N=XX | ľ | N=XX | I | N=XX | ľ | N=XX | ľ | N=XX |
| | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) |
| All Serious Adverse Events | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each System Organ Class | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each Preferred Term | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |

<sup>[1]</sup> Events reported as adjudicated or by site if not adjudicated

<sup>[2]</sup> Denominators of time points are subjects past the visit window or with an event

| | | I | Listing 12 | | | |
|---|---|---|---|---|---|---|
| | Summary of Serious Adverse Events by SOC and PT | | | | | |
| Subject ID | Adverse Event SOC Days Post Any Adverse Any Serious | | | | | |
| XX-XXX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Device-Rel | Table 13 Device-Related Treatment Emergent Adverse Events Summary by System Organ Class and Preferred Term [1] [2] | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Safety Population | | | | | | | | | | |
| After Treatment Prior to Day 30 Prior to Day 30 Prior to Day 60 Prior to Day 60 Prior to Day 90 Prior to Day 9 | | | | | | | | | | |
| | ľ | N=XX | N=XX | | N=XX | | N=XX | | N=XX | |
| | #<br>Events | Subjects<br>w/Event<br>% (n/N) | w/Event # w/Event | | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) |
| All Device-related AEs | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each System Organ Class | | | | | | | | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each Preferred Term | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |

<sup>[1]</sup> Events reported as adjudicated or by site if not adjudicated

<sup>[2]</sup> Denominators of time points are subjects past the visit window or with an event

| | Listing 13 | | | | | |
|---|---|---|---|---|---|---|
| | Summary of Adverse Events Related to Study Treatment | | | | | |
| Subject ID | Adverse Event<br>Number | SOC<br>(Preferred Term) | Days Post<br>Procedure | Any Adverse<br>Event | Any Serious<br>Adverse<br>Event | Event Related to Study Treatment |
| XX-XXX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Device-Related Tr | eatment E | Emergent Serio | ous Advers | Table 14<br>se Events Sumi | mary by S | ystem Organ ( | Class and I | Preferred Teri | m [1] [2] | |
|---|---|---|---|---|---|---|---|---|---|---|
| Safety Population | | | | | | | | | | |
| | Prior | After Treatment Prior to Day 30 Up to Day 60 Up to Day 90 After Day 90 | | After Day 90,<br>up to day 180 | | Total | | | | |
| | 1 | N=XX N=XX | | 1 | N=XX | Γ | N=XX | | N=XX | |
| | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) |
| All Device-related, Serious AEs | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each System Organ Class | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each Preferred Term | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |

<sup>[1]</sup> Events reported as adjudicated or by site if not adjudicated

<sup>[2]</sup> Denominators of time points are subjects past the visit window or with an event

| | Listing 14 | | | | | | |
|---|---|---|---|---|---|---|---|
| | | | Summary of Serious Advers | e Events Related | d to Study Treat | ment | |
| | Subject ID | Adverse Event<br>Number | SOC<br>(Preferred Term) | Days Post<br>Procedure | Any Adverse<br>Event | Any Serious<br>Adverse<br>Event | Event Related to Study Treatment |
| ſ | XX-XXX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Treatment Eme | rgent Adver | se Events Lea | ding to W | Table 15 | | System Organ | Class and | l Preferred Te | erm[1] [2] | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Safety Popula | ation | | | | | |
| | | fter Treatment After Day 30, After Day 60, After Day 90, rior to Day 30 up to Day 60 up to Day 90 up to day 180 | | | , | Total | | | | |
| | ľ | N=XX | ľ | N=XX | | N=XX | N=XX | | N=XX | |
| | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) | #<br>Events | Subjects<br>w/Event<br>% (n/N) |
| All Adverse Events | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each System Organ Class | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |
| each Preferred Term | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) | XX | XX.X<br>(X/XX) |

<sup>[1]</sup> Events reported as adjudicated or by site if not adjudicated

<sup>[2]</sup> Denominators of time points are subjects past the visit window or with an event

| | Listing 15 | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary of Adverse Events Leading to Withdrawal | | | | | | | |
| Subject Adverse Event SOC Days Post Any Adverse Any Serious Event Related to Study Event Led to Subject | | | | | | | Comments | |
| XX-XXX | XX | XX | XX | XX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 16<br>Numerical Rating Scale (NRS) | | | | |
|---|---|---|---|---|
| | Safety Population | | | |
| | Day 30 | Day 60 [1] | Day 90 | Day 180 |
| | N=XX | N=XX | N=XX | N=XX |
| NRS | | | | |
| $Mean \pm SD (N)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX.X, XX.X) | XX.X (XX.X, XX.X) | XX.X (XX.X, XX.X) | XX.X (XX.X, XX.X) |
| Change in NRS from Day 30 | ) | | | |
| $Mean \pm SD (N)$ | N/A | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | N/A | XX.X (XX.X, XX.X) | XX.X (XX.X, XX.X) | XX.X (XX.X, XX.X) |
| Change in NRS from Day 90 | | | | |
| $Mean \pm SD(N)$ | N/A | N/A | N/A | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | N/A | N/A | N/A | XX.X (XX.X, XX.X) |

<sup>[1] 30</sup> subjects in sequential order of enrollment chosen for 60 day visit.

| Listing 16 | | | | |
|---|---|---|---|---|
| Numerical Rating Scale (NRS) | | | | |
| Subject ID | Day 30 | Day 60 | Day 90 | Day 180 |
| XX-XXX | XX | XX | XX | XX |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift

| Table 17 Protocol Deviations ITT Population | | | | |
|---|---|---|---|---|
| | | | N=XX Number of Subje | |
| Category | Reason | Time Period | # Deviations | with Deviation<br>% (n/N) |
| | | Enrollment | XX | XX.X (X/XX) |
| | | Baseline | XX | XX.X (X/XX) |
| | | Treatment | XX | XX.X (X/XX) |
| | | 30 day follow-up | XX | XX.X (X/XX) |
| | | 90 day follow-up | XX | XX.X (X/XX) |
| | | 180 day follow-up | XX | XX.X (X/XX) |
| | | | XX | XX.X (X/XX) |
| | | | XX | XX.X (X/XX) |
| | | | XX | XX.X (X/XX) |
| | | | XX | XX.X (X/XX) |

| | Listing 17 |
|---|---|
| | Protocol Deviations |
| Subject ID | Subject ID Category Reason Time Period |
| XX-XXX XX XX XX | |

Protocol: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental

Lift


| Table 18<br>Study Exit<br>ITT Population | |
|------------------------------------------|----------------------|
| | N=XX |
| Study status, % (n/N) | |
| Complete | XX.X (X/XX) |
| Early exit | XX.X (X/XX) |
| Time to early exit (days) | |
| $Mean \pm SD (N)$ | $XX.X \pm XX.X (XX)$ |
| Median (Min, Max) | XX.X (XX.X, XX.X) |
| Reason for early exit, % (n/N) | |
| Subject withdrew consent [1] | XX.X (X/XX) |
| Study terminated prematurely by sponsor | XX.X (X/XX) |
| Subject non-compliance | XX.X (X/XX) |
| Adverse Event/Serious Adverse Event [2] | XX.X (X/XX) |
| Other [3] | XX.X (X/XX) |

Note: Percentages are based on the number of subjects in the ITT Population.

- [1] See supporting listing for reasons for consent withdrawal
- [2] See supporting listing for adverse events/serious adverse events
- [3] See supporting listing for other reason for early exit

| Listing 18<br>Study Exit | | | | |
|---|---|---|---|---|
| Subject ID | Study Status | Time to Exit (Days) | Reason for Early<br>Exit | Comments |
| XX-XXX | XX | XX | XX | XX |